CLINICAL TRIAL: NCT04888247
Title: HighLife TSMVR Feasibility Study of the Open Cell CLARITY Valve in Patients With Moderate-severe or Severe MR, High Surgical Risk and With a High Risk for Left Ventricular Outflow Tract Obstruction (LVOTO)
Brief Title: HighFLO Study - HighLife Trans-septal Mitral Valve Replacement (TSMVR) Feasibility Study of the Open Cell CLARITY Valve
Acronym: HighFLO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HighLife SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HL-2021-01
Record Dates: First submitted 2021-05-04; First posted 2021-05-17 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Trans-septal mitral valve replacement
  Interventions: Device: CLARITY

INTERVENTIONS:
Device: CLARITY — Trans-septal mitral valve replacement

SUMMARY:
Feasibility, safety and performance of the HighLife CLARITY TSMV and its delivery system

DETAILED DESCRIPTION:
Study to assess the feasibility, safety, and performance of the HighLife CLARITY TSMV, and its deliver systems, in NYHA Class ≥ II-IV patients with moderate-severe or severe mitral regurgitation who are at high risk for surgical treatment according to the local multidisciplinary Heart Team decision, and who are at high risk for potential LVOT obstruction(LVOTO).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Moderate-severe or severe mitral regurgitation (≥ 3+)
3. Patient has New York Heart Association (NYHA) Functional Class II, III or ambulatory IV
4. Patient is under guideline directed medical therapy for at least one month, as reviewed and confirmed by the local multidisciplinary Heart Team
5. Patient is high-risk for open-heart surgery based on the assessment of the multidisciplinary Heart Team using standard scoring systems and consideration of co-morbidities, frailty, and disability
6. Patient meets the anatomical criteria for HighLife valve
7. Patient is willing to participate in the study and provides signed informed consent
8. Patients with a high risk for LVOTO

Exclusion Criteria:

1. Any stroke/TIA within 30 days
2. Severe symptomatic carotid stenosis (> 70% by non-invasive imaging)
3. Active infections requiring antibiotic therapy
4. Active ulcer or gastro-intestinal bleeding in the past 3 months
5. History of bleeding diathesis, coagulopathy or refusal of future blood transfusion
6. Patients in whom TEE is not feasible
7. Patients who are pregnant or lactating, or plan to get pregnant in the next 12 months.
8. Patient is unable to comply with the follow-up schedule and assessments
9. Participation in another clinical investigation at the time of inclusion
10. Patient has known allergies to the device components or contrast medium
11. Patient cannot tolerate anticoagulation or antiplatelet therapy
12. Patients with a life expectancy of less than 12 months due to non-cardiac conditions
13. Patient had permanent pacemaker, or similar device with implantable cardiac leads (i.e. resynchronization therapy) within the last 3 months

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2031-02-01 (Estimated)

PRIMARY OUTCOMES:
Rate of subjects meeting Technical Success | 24 hours
  * Successful vascular access, delivery and retrieval of the HighLife delivery systems
  * Deployment and correct positioning of the HighLife 28mm CLARITY TSMV
  * Freedom from additional emergency surgery or re-intervention related to the device or access procedure, that occurred (was initiated) during the procedure. Any emergency surgery or re-intervention that occurs after the patient exits the procedure room/cath lab in stable condition will be captured as an AE/SAE
  * Successful vascular access, delivery and retrieval of the HighLife delivery systems
  * Deployment and correct positioning of the HighLife 28mm CLARITY TSMV
  * Freedom from additional emergency surgery or re-intervention related to the device or access procedure, that occurred (was initiated) during the procedure. Any emergency surgery or re-intervention that occurs after the patient exits the procedure room/cath lab in stable condition will be captured as an AE/SAE

CONTACTS AND LOCATIONS:
Locations (14):
- Australia (3):
  - Wesley Hospital, Auchenflower
  - Mount Hospital, Perth
  - Macquarie University Hospital, Sydney
- Belgium (2):
  - AZ St. Jan - Brugge, Bruges
  - UZ Leuven, Leuven
- France (4):
  - CHU Lille, Lille
  - Centre Hospitalo - Univ de Nantes, Nantes
  - CHU de Rennes, Rennes
  - Cliniue Pasteur, Toulouse
- Germany (2):
  - Deutsches Herzzentrum Munchen, Munich
  - University Hospital Ulm, Ulm
- Poland (2):
  - Medical University of Silesia, Katowice
  - Medical University of Warsaw, Warsaw
- Brighton and Sussex University Hospital, Brighton, United Kingdom